CLINICAL TRIAL: NCT01383421
Title: A Post-Marketing Observational Study (PMOS) to Determine the Effectiveness and Patient Satisfaction With Adalimumab Treatment in Patients With Rheumatoid Arthritis (PASSION Study)
Brief Title: Observational Study to Explore the Effectiveness of Adalimumab Treatment in Conjunction With Utilization of a Patient Support Program (PSP)
Acronym: PASSION
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-072
Record Dates: First submitted 2011-06-26; First posted 2011-06-28 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Patient Support Program; adalimumab
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants With RA Receiving Adalimumab: Participants with RA who were prescribed adalimumab based on current clinical practice criteria (regardless of participation in the study), with the first dose corresponding to the Enrollment/Baseline visit.
  All participants were offered to participate in the PSP while treated with ADA for their RA.

SUMMARY:
This study is a non-confirmatory post-marketing observational study to explore and describe the effectiveness of adalimumab on rheumatoid arthritis (RA) treatment course and participant satisfaction over time in context with utilization of a patient support program (PSP). The core elements of the PSP were call centers (in and outbound)/hotlines, nursing services, starter packs, provision of educational materials (print and digital) regarding RA and adalimumab, and injection guides. Other elements of the PSP, which varied between countries, included (but were not limited to) refill reminders, email contacts, support groups, and newsletters.

DETAILED DESCRIPTION:
The main objectives of the study are to examine the effectiveness of adalimumab treatment with respect to PSPs by means of Health Assessment Questionnaire Disability Index (HAQ-DI), Disease Activity Score (DAS28) results, and European League Against Rheumatism (EULAR) response criteria, as well as to evaluate the contribution of PSP to disease control, treatment continuation over time, participant's satisfaction, and PSP utilization.

The primary endpoint is the percentage of participants achieving a minimal clinically important difference (MCID) in HAQ-DI at Week 78. (MCID is improvement of at least 0.22 in HAQ-DI compared to Baseline). Secondary endpoints include the percentage of participants achieving MCID in HAQ-DI at Weeks 12, 24, 36, 52, 64 and other effectiveness parameters, including: changes in DAS28, Simplified Disease Activity Index (SDAI), Clinical Disease Activity Index (CDAI), ACR 20/50/70 and EULAR moderate and good responses. Other secondary endpoints include health outcomes assessments including HAQ-DI, Work Productivity and Activity Impairment (WPAI), Compliance Questionnaire Rheumatology (CQR), and Treatment Satisfaction Questionnaire for Medication (TSQM) scores, expectation regarding PSP and health management via Patient Activation Measure (PAM-13), change in participant perceptions as measured by the Beliefs about Medicines Questionnaire (BMQ), and satisfaction with PSP as measured by PSP satisfaction assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged at least 18 years that has been newly prescribed adalimumab therapy according to the local product label, with the first dose corresponding to the Enrollment/Baseline visit.
* Patient with a diagnosis of moderate to severe RA, who has had insufficient response to one or more disease-modifying antirheumatic drugs (DMARDs), and has a prescription of adalimumab according to the local regulations.
* Patients should be evaluated for tuberculosis (TB) exposure/risk factors for active and latent TB (per local requirements and according to the local product label).
* Patients must be able and willing to provide written authorization to disclose and use personal health information (and informed consent where applicable) and comply with the requirements of this study protocol as well as agree to data being collected and provided to AbbVie.

Exclusion Criteria:

* Patients should not be enrolled if they cannot be treated in accordance with the local adalimumab product label.
* Patients treated with > 1 prior biologic DMARD for RA. Any prior treatment with adalimumab is prohibited.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Representative disease population selected from rheumatology clinics in the countries selected.
Sampling Method: Non-Probability Sample
Enrollment: 1036 (Actual)
Dates: Start 2011-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmina Kalabic, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Van den Bosch F, Ostor AJK, Wassenberg S, Chen N, Wang C, Garg V, Kalabic J. Impact of Participation in the Adalimumab (Humira) Patient Support Program on Rheumatoid Arthritis Treatment Course: Results from the PASSION Study. Rheumatol Ther. 2017 Jun;4(1):85-96. doi: 10.1007/s40744-017-0061-7. Epub 2017 Mar 30. PMID 28361468
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With RA Receiving Adalimumab: Participants with RA who initiated adalimumab based on current clinical practice criteria (regardless of participation in the study), with the first dose corresponding to the Enrollment/Baseline visit.
  All participants were offered to participate in the PSP while treated by ADA for their RA.
Period: Overall Study
Arm/Group | Participants With RA Receiving Adalimumab
Started | 1025 (ITT population: all enrolled participants who received at least 1 dose of study drug.)
Completed | 679
Not Completed | 346

BASELINE CHARACTERISTICS:
Population: ITT population: all enrolled participants who received at least 1 dose of study drug.
Groups:
- Participants With RA Receiving Adalimumab: Participants with RA who initiated adalimumab based on current clinical practice criteria (without taking participation in the study into account), with the first dose corresponding to the Enrollment/Baseline visit.
  All participants were offered to participate in the PSP while treated by ADA for their RA.
Arm/Group | Participants With RA Receiving Adalimumab
Number analyzed (Participants) | 1025
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (13.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 790
  Male | 235

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Minimal Clinically Important Difference (MCID) in the Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 78
Description: The HAQ-DI is a self-reported assessment of how the participant's illness affects their ability to function in their daily life over the past week. The HAQ-DI for a participant is calculated as the mean of the following 8 category scores (range: 0 to 3): Dressing and Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. A lower score demonstrates less disability. The MCID in HAQ-DI was defined as an improvement of at least 0.22 in HAQ-DI compared to Baseline.
Time Frame: Baseline, Week 78
Population: Intent to treat analysis population: all enrolled participants who received at least 1 dose of adalimumab. Non-responder imputation.
Measure: Number; unit: percentage of participants
Groups:
- Participants With RA Receiving Adalimumab: PSP User: Participants with RA who initiated adalimumab based on current clinical practice criteria (regardless of participation in the study), with the first dose corresponding to the Enrollment/Baseline visit.
  These participants utilized the PSP that was offered.
- Participants With RA Receiving Adalimumab: PSP Non-User: Participants with RA who initiated adalimumab based on current clinical practice criteria (regardless of participation in the study), with the first dose corresponding to the Enrollment/Baseline visit.
  These participants did not utilize the PSP that was offered.
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 499 | 526
percentage of participants | 48.1 | 37.8
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Test type: Superiority; p < 0.001, Chi-squared — Statistical significance was set at P = 0.05

2. Secondary Outcome: Percentage of Participants Achieving a MCID in the HAQ-DI at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 499 | 526
percentage of participants | 60.9 [56.6 to 65.2] | 50.0 [45.7 to 54.3]

3. Secondary Outcome: Percentage of Participants Achieving a MCID in the HAQ-DI at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 499 | 526
percentage of participants | 52.3 [47.9 to 56.7] | 46.4 [42.1 to 50.6]
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Test type: Superiority; p = 0.058, Chi-squared — Statistical significance was set at P = 0.05

4. Secondary Outcome: Percentage of Participants Achieving a MCID in the HAQ-DI at Week 36
Description: as for outcome 1
Time Frame: Baseline, Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 499 | 526
percentage of participants | 49.9 [45.5 to 54.3] | 43.0 [38.7 to 47.2]

5. Secondary Outcome: Percentage of Participants Achieving a MCID in the HAQ-DI at Week 52
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 499 | 526
percentage of participants | 48.5 [44.1 to 52.9] | 39.2 [35.0 to 43.3]
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Test type: Superiority; p = 0.003, Chi-squared — Statistical significance was set at P = 0.05

6. Secondary Outcome: Percentage of Participants Achieving a MCID in the HAQ-DI at Week 64
Description: as for outcome 1
Time Frame: Baseline, Week 64
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 499 | 526
percentage of participants | 48.3 [43.9 to 52.7] | 37.3 [33.1 to 41.4]

7. Other Pre Specified Outcome: Mean Change From Baseline in With 28-Joint Disease Activity Score of C-reactive Protein (DAS28[CRP]) at Weeks 24, 52, and 78
Description: The DAS28 is a validated combined index of RA disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher numbers indicating more disease activity.
Time Frame: Baseline and Weeks 24, 52, 78
Population: Intent to treat analysis population: all enrolled participants who received at least 1 dose of adalimumab and had an assessment at given time point. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Participants With RA Receiving Adalimumab: Participants with RA who initiated adalimumab based on current clinical practice criteria (regardless of participation in the study), with the first dose corresponding to the Enrollment/Baseline visit.
  All participants were offered to participate in the PSP while treated with ADA for their RA.
Arm/Group | Participants With RA Receiving Adalimumab | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 852 | 427 | 425
units on a scale
  Change at Week 24: number analyzed (Participants) | 822 | 412 | 410
  Change at Week 24 | -2.09 (1.48) | -2.24 (1.55) | -1.94 (1.39)
  Change at Week 52: number analyzed (Participants) | 848 | 425 | 423
  Change at Week 52 | -2.11 (1.56) | -2.31 (1.62) | -1.92 (1.49)
  Change at Week 78 | -2.15 (1.63) | -2.33 (1.68) | -1.97 (1.56)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 24; Test type: Superiority; p = 0.027, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -0.203, Standard Error of Mean 0.092
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 52; Test type: Superiority; p = 0.006, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -0.260, Standard Error of Mean 0.094
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 78; Test type: Superiority; p = 0.018, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -0.233, Standard Error of Mean 0.098

8. Other Pre Specified Outcome: Mean Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 24, 52, and 78
Description: The SDAI is a validated measure of RA disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global disease activity assessed by the participant on a visual analogue scale from 0 to 10 (cm) , global disease activity assessed by an investigator on a visual analogue scale from 0 to 10 (cm), and serum levels of C-reactive protein (mg/dL) were included in the SDAI score. Scores on the SDAI range from 0 to 86. An SDAI score ≥26.1 indicates high disease activity, an SDAI score between 11.1 and 26.0 indicates moderate disease activity, an SDAI score between 3.4 and 11.0 indicates low disease activity, and an SDAI score ≤3.3 indicates clinical remission.
Time Frame: Baseline, Weeks 24, 52, and 78
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 831 | 411 | 420
units on a scale
  Change at Week 24: number analyzed (Participants) | 803 | 399 | 404
  Change at Week 24 | -21.78 (16.42) | -23.59 (17.62) | -20.00 (14.95)
  Change at Week 52: number analyzed (Participants) | 827 | 409 | 418
  Change at Week 52 | -21.97 (17.01) | -24.46 (17.88) | -19.54 (15.77)
  Change at Week 78 | -22.12 (17.70) | -24.50 (18.49) | -19.80 (16.58)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 24; Test type: Superiority; p = 0.059, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -1.686, Standard Error of Mean 0.893
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 52; Test type: Superiority; p = 0.003, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -2.697, Standard Error of Mean 0.903
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 78; Test type: Superiority; p = 0.010, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -2.447, Standard Error of Mean 0.945

9. Other Pre Specified Outcome: Mean Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 24, 52, and 78
Description: The CDAI is a validated measure of RA disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global health assessed by the participant on a visual analogue scale from 0 to 10 (cm), and global health assessed by an investigator on a visual analogue scale from 0 to 10 (cm) were included in the CDAI score. Scores on the CDAI range from 0 to 76. A CDAI score ≥22.1 indicates high disease activity, a CDAI score between 10.1 and 22.0 indicates moderate disease activity, a CDAI score between 2.9 and 10.0 indicates low disease activity, and a CDAI score ≤2.8 indicates clinical remission.
Time Frame: Baseline, Weeks 24, 52, and 78
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 893 | 438 | 455
units on a scale
  Change at Week 24: number analyzed (Participants) | 880 | 435 | 445
  Change at Week 24 | -20.42 (15.16) | -21.94 (15.60) | -18.93 (14.58)
  Change at Week 52: number analyzed (Participants) | 890 | 438 | 452
  Change at Week 52 | -20.61 (15.63) | -22.58 (15.84) | -18.71 (15.21)
  Change at Week 78 | -20.56 (16.52) | -22.66 (16.67) | -18.55 (16.13)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 24; Test type: Superiority; p = 0.023, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -1.791, Standard Error of Mean 0.788
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 52; Test type: Superiority; p = 0.002, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -2.549, Standard Error of Mean 0.818
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 78; Test type: Superiority; p = 0.002, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -2.734, Standard Error of Mean 0.872

10. Other Pre Specified Outcome: Percentage of Participants Achieving American College of Rheumatology 20%, 50%, 70% (ACR20, ACR50, ACR70) Response at Week 78
Description: ACR20/50/70 response is a 20%/50%/70% improvement in a participant's disease condition compared to Baseline. A participant is considered an ACR20/50/70 responder if the following 3 criteria are met: ≥ 20/50/70% improvement in 28 tender joint count; ≥ 20/50/70% improvement in swollen joint count; ≥ 20/50/70% improvement in at least 3 of the following 5 assessments:
  * Patient's assessment of pain
  * Patient's global assessment of disease activity
  * Physician's global assessment of disease activity
  * HAQ-DI
  * Acute phase reactant value (CRP or erythrocyte sedimentation date [ESR])
Time Frame: Week 78
Population: Intent to treat analysis population: all enrolled participants who received at least 1 dose of adalimumab and had non-missing visit values. Observed cases.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 316 | 274
percentage of participants
  ACR20 | 75.9 | 72.6
  ACR50 | 58.5 | 50.4
  ACR70 | 38.6 | 32.5

11. Other Pre Specified Outcome: Percentage of Participants With a Good or Moderate European League Against Rheumatism (EULAR) Response (Using DAS28[ESR] at Week 78
Description: A EULAR response reflects improvement in disease activity and attainment of a lower degree of disease activity based on the DAS28(ESR) score. The DAS28(ESR) score ranges from 0-10, with higher scores indicating more disease activity.
  * A Good Response is defined as an improvement (decrease) in the DAS28 of > 1.2 compared with Baseline and attainment of a DAS28 score of ≤ 3.2.
  * A Moderate Response is defined as either: an improvement (decrease) in the DAS28 of > 0.6 and ≤ 1.2 from Baseline and attainment of a DAS28 score of ≤ 5.1; or, an improvement (decrease) in the DAS28 of > 1.2 from Baseline and attainment of a DAS28 score of > 3.2.
  * No Response is defined as either an improvement (decrease) in the DAS28 of ≤ 0.6, or an improvement (decrease) in the DAS28 of > 0.6 and ≤ 1.2 and attainment of a DAS28 of > 5.1
Time Frame: Week 78
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 268 | 208
percentage of participants
  Good | 58.6 | 59.1
  Moderate | 28.4 | 31.3
  No Response | 13.1 | 9.6

12. Other Pre Specified Outcome: Percentage of Participants With a Good or Moderate EULAR Response (Using DAS28[CRP] at Week 78
Description: A EULAR response reflects improvement in disease activity and attainment of a lower degree of disease activity based on the DAS28(CRP) score. The DAS28(CRP) score ranges from 0-10, with higher scores indicating more disease activity.
  * A Good Response is defined as an improvement (decrease) in the DAS28 of >1.2 compared with Baseline and attainment of a DAS28 score of ≤ 3.2.
  * A Moderate Response is defined as either: an improvement (decrease) in the DAS28 of > 0.6 and ≤ 1.2 from Baseline and attainment of a DAS28 score of ≤ 5.1; or, an improvement (decrease) in the DAS28 of > 1.2 from Baseline and attainment of a DAS28 score of > 3.2.
  * No Response is defined as either an improvement (decrease) in the DAS28 of ≤ 0.6, or an improvement (decrease) in the DAS28 of > 0.6 and ≤ 1.2 and attainment of a DAS28 of > 5.1
Time Frame: Week 78
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 275 | 237
percentage of participants
  Good | 65.1 | 70.9
  Moderate | 22.9 | 19.8
  None | 12.0 | 9.3

13. Other Pre Specified Outcome: Mean Change From Baseline in Work Productivity and Activity Impairment (WPAI) at Week 24
Description: The WPAI assessed impact of RA on work productivity and non-work activity limitation. Participants were asked during the past 7 days: how many hours did you miss from work because of problems associated with RA (absenteeism), how many hours did you miss from work because of any other reason, such as vacation, holidays, time off to participate in this study (presenteeism), how much did your RA affect your productivity while you were working (overall work impairment), and much did RA affect your ability to do your regular daily activities, other than work at a job (activity impairment). Answers were rated on an 11-point scale, with 0 indicating "RA had no effect on this" and 10 indicating "RA completely prevented me from this." A decrease in the WPAI score indicates improvement.
Time Frame: Baseline, Week 24
Population: Intent to treat analysis population: all enrolled participants who received at least 1 dose of adalimumab and had an assessment. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 932 | 474 | 458
units on a scale
  WPAI absenteeism: number analyzed (Participants) | 287 | 149 | 138
  WPAI absenteeism | -3.81 (29.07) | -2.32 (25.40) | -5.43 (32.58)
  WPAI presenteeism: number analyzed (Participants) | 330 | 167 | 163
  WPAI presenteeism | -17.88 (27.75) | -18.68 (27.41) | -17.06 (28.15)
  WPAI overall work impairment: number analyzed (Participants) | 285 | 148 | 137
  WPAI overall work impairment | -17.85 (31.74) | -17.55 (31.79) | -18.17 (31.80)
  WPAI activity impairment | -22.04 (27.49) | -23.90 (29.03) | -20.11 (25.69)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI absenteeism; Test type: Superiority; p = 0.625, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 1.333, Standard Error of Mean 2.725
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI presenteeism; Test type: Superiority; p = 0.736, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -0.824, Standard Error of Mean 2.441
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI overall work impairment; Test type: Superiority; p = 0.700, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 1.207, Standard Error of Mean 3.126
Statistical Analysis 4: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI activity impairment; Test type: Superiority; p = 0.023, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -3.552, Standard Error of Mean 1.561

14. Other Pre Specified Outcome: Mean Change From Baseline in WPAI at Week 52
Description: as for outcome 13
Time Frame: Baseline, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 944 | 478 | 466
units on a scale
  WPAI absenteeism: number analyzed (Participants) | 299 | 152 | 147
  WPAI absenteeism | -3.97 (30.75) | -2.80 (29.25) | -5.18 (32.28)
  WPAI presenteeism: number analyzed (Participants) | 337 | 169 | 168
  WPAI presenteeism | -17.69 (28.23) | -18.34 (26.56) | -17.02 (29.88)
  WPAI overall work impairment: number analyzed (Participants) | 299 | 152 | 147
  WPAI overall work impairment | -17.24 (33.21) | -17.77 (32.09) | -16.69 (34.44)
  WPAI activity impairment | -23.04 (28.63) | -25.06 (29.23) | -20.97 (27.89)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI absenteeism; Test type: Superiority; p = 0.890, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 0.380, Standard Error of Mean 2.736
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI presenteeism; Test type: Superiority; p = 0.835, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -0.527, Standard Error of Mean 2.523
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI overall work impairment; Test type: Superiority; p = 0.883, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -0.471, Standard Error of Mean 3.205
Statistical Analysis 4: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI activity impairment; Test type: Superiority; p = 0.019, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -3.792, Standard Error of Mean 1.611

15. Other Pre Specified Outcome: Mean Change From Baseline in WPAI at Week 78
Description: as for outcome 13
Time Frame: Baseline, Week 78
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 946 | 478 | 468
units on a scale
  WPAI absenteeism: number analyzed (Participants) | 307 | 156 | 151
  WPAI absenteeism | -6.92 (29.92) | -5.71 (27.55) | -8.17 (32.23)
  WPAI presenteeism: number analyzed (Participants) | 345 | 172 | 173
  WPAI presenteeism | -18.41 (29.43) | -19.07 (28.19) | -17.75 (30.69)
  WPAI overall work impairment: number analyzed (Participants) | 307 | 156 | 151
  WPAI overall work impairment | -21.13 (33.33) | -22.28 (30.70) | -19.94 (35.90)
  WPAI activity impairment | -23.52 (29.41) | -26.42 (29.28) | -20.56 (29.28)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI absenteeism; Test type: Superiority; p = 0.873, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -0.409, Standard Error of Mean 2.548
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI presenteeism; Test type: Superiority; p = 0.753, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -0.817, Standard Error of Mean 2.598
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI overall work impairment; Test type: Superiority; p = 0.461, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -2.334, Standard Error of Mean 3.159
Statistical Analysis 4: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; WPAI activity impairment; Test type: Superiority; p < 0.001, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = -5.537, Standard Error of Mean 1.624

16. Other Pre Specified Outcome: Mean Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) Scores at Week 24
Description: TSQM is a 14-point measure to show that adherence is expected to be related with participants' satisfaction with therapy and such satisfaction can be a function of not only the effect of the treatment, but also the services offered. TSQM responses are used to derive scores for scales measuring effectiveness, side effects, convenience, and global satisfaction (based on participant evaluation over the last 2 to 3 weeks, or since last medication use). Scores for each of the 4 scales range from 0 to 100 with higher scores indicating a better state or outcome (e.g., greater perceived effectiveness or satisfaction).
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 656 | 387 | 269
units on a scale
  TSQM convenience | 5.51 (20.02) | 6.67 (20.27) | 3.85 (19.58)
  TSQM effectiveness: number analyzed (Participants) | 630 | 368 | 262
  TSQM effectiveness | 14.45 (31.12) | 14.56 (32.25) | 14.29 (29.53)
  TSQM global satisfaction: number analyzed (Participants) | 650 | 383 | 267
  TSQM global satisfaction | 11.20 (26.90) | 11.44 (26.43) | 10.85 (27.60)
  TSQM side effects: number analyzed (Participants) | 613 | 367 | 246
  TSQM side effects | 8.17 (32.05) | 8.21 (30.91) | 8.10 (33.74)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM convenience; Test type: Superiority; p = 0.017, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 2.973, Standard Error of Mean 1.245
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM effectiveness; Test type: Superiority; p = 0.164, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 2.843, Standard Error of Mean 2.042
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM global satisfaction; Test type: Superiority; p = 0.003, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 5.473, Standard Error of Mean 1.866
Statistical Analysis 4: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM side effects; Test type: Superiority; p = 0.335, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 1.705, Standard Error of Mean 1.769

17. Other Pre Specified Outcome: Mean Change From Baseline in TSQM Scores at Week 52
Description: as for outcome 16
Time Frame: Baseline, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 705 | 413 | 292
units on a scale
  TSQM convenience | 6.30 (20.15) | 7.38 (19.94) | 4.77 (20.38)
  TSQM effectiveness | 15.79 (30.80) | 16.06 (31.84) | 15.41 (29.38)
  TSQM global satisfaction | 11.94 (26.68) | 12.53 (26.35) | 11.12 (27.15)
  TSQM side effects | 8.28 (32.29) | 8.09 (31.23) | 8.55 (33.81)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM convenience; Test type: Superiority; p = 0.021, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 2.728, Standard Error of Mean 1.183
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM effectiveness; Test type: Superiority; p = 0.106, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 3.124, Standard Error of Mean 1.930
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM global satisfaction; Test type: Superiority; p = 0.002, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 5.572, Standard Error of Mean 1.756
Statistical Analysis 4: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM side effects; Test type: Superiority; p = 0.269, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 1.885, Standard Error of Mean 1.704

18. Other Pre Specified Outcome: Mean Change From Baseline in TSQM Scores at Week 78
Description: as for outcome 16
Time Frame: Baseline, Week 78
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 722 | 422 | 300
units on a scale
  TSQM convenience | 6.20 (20.14) | 7.23 (19.87) | 4.76 (20.47)
  TSQM effectiveness: number analyzed (Participants) | 695 | 401 | 294
  TSQM effectiveness | 15.14 (30.58) | 16.24 (31.22) | 13.62 (29.68)
  TSQM global satisfaction: number analyzed (Participants) | 717 | 417 | 300
  TSQM global satisfaction | 10.93 (27.07) | 11.68 (26.67) | 9.87 (27.63)
  TSQM side effects: number analyzed (Participants) | 687 | 403 | 284
  TSQM side effects | 8.32 (31.72) | 8.37 (30.98) | 8.25 (32.80)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM convenience; Test type: Superiority; p = 0.049, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 2.324, Standard Error of Mean 1.177
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM effectiveness; Test type: Superiority; p = 0.011, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 4.929, Standard Error of Mean 1.929
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM global satisfaction; Test type: Superiority; p < 0.001, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 5.997, Standard Error of Mean 1.775
Statistical Analysis 4: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; TSQM side effects; Test type: Superiority; p = 0.272, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 1.823, Standard Error of Mean 1.657

19. Other Pre Specified Outcome: Mean Change From Baseline in Compliance Questionnaire Rheumatology (CQR) at Weeks 24, 52, and 78
Description: The CQR includes 19 items and measures RA treatment-specific compliance/adherence. Participants select an answer based on whether they agree with each statement. The agreements are based on a 4-point Likert scale with anchors "don't agree at all" (score = 1), "don't agree" (score = 2), "agree" (score = 3), and "agree very much" (score = 4). The total score is calculated by summing all 19 items and subtracting 19 from the total and dividing by 0.57. The compliance score ranges between 0 (complete non-compliance) to 100 (perfect compliance).
Time Frame: Baseline, Week 24, 52, and 78
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 957 | 490 | 467
units on a scale
  Change at Week 24: number analyzed (Participants) | 946 | 488 | 458
  Change at Week 24 | 2.23 (10.11) | 2.44 (9.78) | 2.01 (10.45)
  Change at Week 52: number analyzed (Participants) | 956 | 490 | 466
  Change at Week 52 | 2.20 (10.75) | 2.39 (10.20) | 1.99 (11.30)
  Change at Week 78 | 2.06 (10.53) | 2.30 (9.63) | 1.80 (11.41)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 24; Test type: Superiority; p = 0.154, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 0.817, Standard Error of Mean 0.572
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 52; Test type: Superiority; p = 0.198, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 0.772, Standard Error of Mean 0.599
Statistical Analysis 3: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Week 78; Test type: Superiority; p = 0.131, ANCOVA — Statistical significance was set at P = 0.05; LS mean difference and P value are from ANCOVA model adjusting for corresponding Baseline values; LS Mean Difference = 0.884, Standard Error of Mean 0.585

20. Other Pre Specified Outcome: Percentage of Participants Who Demonstrated Improvement From Baseline or Who Remained at Level 4 From Baseline on the Patient Activation Measure (PAM-13) at Week 78
Description: The PAM-13 is a measure used to assess the participant's knowledge, skill, and confidence for self-management of his/her health. Participants are given a questionnaire of 13 statements to which they responded that they strongly disagree (1), disagree (2), agree (3), or strongly agree (4). Responses are summed and averaged to come up with an overall score of level 1 through level 4, with higher levels indicating more knowledge, skill and confidence for self-management.
Time Frame: Baseline, Week 78
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 499 | 526
percentage of participants | 35.7 | 28.1

21. Other Pre Specified Outcome: Percentage of Participants Who Started and Remained at Level 4 From Baseline to Week 78 on the PAM-13
Description: as for outcome 20
Time Frame: Baseline, Week 78
Population: Intent to treat analysis population: all enrolled participants who received at least 1 dose of adalimumab and were at Level 4 at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 103 | 83
percentage of participants | 52.4 | 28.9

22. Other Pre Specified Outcome: Percentage of Participants Who Started at Level 3 (or Above) at Baseline and Remained at Level 3 or Improved to Level 4 on the PAM-13 at Week 78
Description: as for outcome 20
Time Frame: Baseline, Week 78
Population: Intent to treat analysis population: all enrolled participants who received at least 1 dose of adalimumab and were at Level 3 or 4 at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 203 | 208
percentage of participants | 64.5 | 53.8

23. Other Pre Specified Outcome: Change From Baseline Means in the Beliefs About Medicines Questionnaire (BMQ) at Week 78
Description: The BMQ consists of 11 questions used to assess the participant's beliefs about medication and the necessity of medications prescribed to them for rheumatoid arthritis. Each question answered from 'strongly disagree' to 'strongly agree,' with some questions attributed to the necessity sub-scale, and others to the concern sub-scale. Each answer is scaled from 1 to 5. The necessity sub-scale is calculated by taking the average of necessity scores, and the concern sub-scale is calculated by taking the average of the concern scores. Higher scores on the necessity sub-scale represent the stronger perceptions of the participant for the necessity of their medication. Similarly, higher scores on the concerns sub-scale represent stronger concerns about the potential negative effects of their medications.
Time Frame: Baseline, Week 78
Population: Intent to treat analysis population: all enrolled participants who received at least 1 dose of adalimumab and had non-missing Baseline and at least 1 non-missing post-Baseline value. Observed cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA Receiving Adalimumab: PSP User | Participants With RA Receiving Adalimumab: PSP Non-User
Number analyzed (Participants) | 409 | 362
units on a scale
  Necessity | -0.03 (0.743) | -0.04 (0.729)
  Concern: number analyzed (Participants) | 409 | 361
  Concern | -0.12 (0.902) | -0.17 (0.842)
Statistical Analysis 1: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Necessity; Test type: Superiority; p = 0.019, ANCOVA — Statistical significance was set at P = 0.05; P value is from an ANCOVA model adjusting for Baseline; LS Mean Between Group Change = 0.100, Standard Error of Mean 0.0429
Statistical Analysis 2: Comparison: Participants With RA Receiving Adalimumab: PSP User vs Participants With RA Receiving Adalimumab: PSP Non-User; Concern; Test type: Superiority; p = 0.560, ANCOVA — Statistical significance was set at P = 0.05; P value is from an ANCOVA model adjusting for Baseline; LS Mean Between Group Change = 0.000, Standard Error of Mean 0.0526

24. Other Pre Specified Outcome: PSP Satisfaction Questionnaire Responses at Week 12
Description: The PSP satisfaction questionnaire evaluates the participant's satisfaction with specific PSP components as well as overall program satisfaction through the participant's selecting the response that best reflects their opinion: 1=very good; 2=good; 3=less satisfying; 4=I do not use the services. The percentage of participants at each response level per question is presented.
Time Frame: Week 12
Population: Intent to treat analysis population: all enrolled participants who received at least 1 dose of adalimumab and had an assessment. Observed cases.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User
Number analyzed (Participants) | 465
percentage of participants
  Relieves my daily burden: score 1: number analyzed (Participants) | 457
  Relieves my daily burden: score 1 | 24.1
  Relieves my daily burden: score 2: number analyzed (Participants) | 457
  Relieves my daily burden: score 2 | 32.6
  Relieves my daily burden: score 3: number analyzed (Participants) | 457
  Relieves my daily burden: score 3 | 14.7
  Relieves my daily burden: score 4: number analyzed (Participants) | 457
  Relieves my daily burden: score 4 | 28.7
  Is always there for me: score 1: number analyzed (Participants) | 455
  Is always there for me: score 1 | 32.5
  Is always there for me: score 2: number analyzed (Participants) | 455
  Is always there for me: score 2 | 39.1
  Is always there for me: score 3: number analyzed (Participants) | 455
  Is always there for me: score 3 | 7.9
  Is always there for me: score 4: number analyzed (Participants) | 455
  Is always there for me: score 4 | 20.4
  Offers real added value service: score 1: number analyzed (Participants) | 454
  Offers real added value service: score 1 | 29.7
  Offers real added value service: score 2: number analyzed (Participants) | 454
  Offers real added value service: score 2 | 38.1
  Offers real added value service: score 3: number analyzed (Participants) | 454
  Offers real added value service: score 3 | 8.6
  Offers real added value service: score 4: number analyzed (Participants) | 454
  Offers real added value service: score 4 | 23.6
  Is exceptional: score 1: number analyzed (Participants) | 452
  Is exceptional: score 1 | 28.1
  Is exceptional: score 2: number analyzed (Participants) | 452
  Is exceptional: score 2 | 40.5
  Is exceptional: score 3: number analyzed (Participants) | 452
  Is exceptional: score 3 | 10.0
  Is exceptional: score 4: number analyzed (Participants) | 452
  Is exceptional: score 4 | 21.5
  PSP in total: score 1: number analyzed (Participants) | 459
  PSP in total: score 1 | 39.0
  PSP in total: score 2: number analyzed (Participants) | 459
  PSP in total: score 2 | 35.9
  PSP in total: score 3: number analyzed (Participants) | 459
  PSP in total: score 3 | 2.0
  PSP in total: score 4: number analyzed (Participants) | 459
  PSP in total: score 4 | 23.1
  Call center/hotline: score 1: number analyzed (Participants) | 458
  Call center/hotline: score 1 | 33.2
  Call center/hotline: score 2: number analyzed (Participants) | 458
  Call center/hotline: score 2 | 23.6
  Call center/hotline: score 3: number analyzed (Participants) | 458
  Call center/hotline: score 3 | 2.0
  Call center/hotline: score 4: number analyzed (Participants) | 458
  Call center/hotline: score 4 | 41.3
  Educational materials about life with RA: score 1: number analyzed (Participants) | 463
  Educational materials about life with RA: score 1 | 41.7
  Educational materials about life with RA: score 2: number analyzed (Participants) | 463
  Educational materials about life with RA: score 2 | 40.2
  Educational materials about life with RA: score 3: number analyzed (Participants) | 463
  Educational materials about life with RA: score 3 | 2.2
  Educational materials about life with RA: score 4: number analyzed (Participants) | 463
  Educational materials about life with RA: score 4 | 16.0
  Educational materials about adalimumab: score 1: number analyzed (Participants) | 461
  Educational materials about adalimumab: score 1 | 40.6
  Educational materials about adalimumab: score 2: number analyzed (Participants) | 461
  Educational materials about adalimumab: score 2 | 41.4
  Educational materials about adalimumab: score 3: number analyzed (Participants) | 461
  Educational materials about adalimumab: score 3 | 1.7
  Educational materials about adalimumab: score 4: number analyzed (Participants) | 461
  Educational materials about adalimumab: score 4 | 16.3
  Injection guide: score 1 | 52.3
  Injection guide: score 2 | 38.5
  Injection guide: score 3 | 0.4
  Injection guide: score 4 | 8.8
  Nursing services: score 1: number analyzed (Participants) | 463
  Nursing services: score 1 | 37.4
  Nursing services: score 2: number analyzed (Participants) | 463
  Nursing services: score 2 | 18.6
  Nursing services: score 3: number analyzed (Participants) | 463
  Nursing services: score 3 | 0.2
  Nursing services: score 4: number analyzed (Participants) | 463
  Nursing services: score 4 | 43.8
  Email contact: score 1: number analyzed (Participants) | 459
  Email contact: score 1 | 9.6
  Email contact: score 2: number analyzed (Participants) | 459
  Email contact: score 2 | 11.8
  Email contact: score 3: number analyzed (Participants) | 459
  Email contact: score 3 | 0.9
  Email contact: score 4: number analyzed (Participants) | 459
  Email contact: score 4 | 77.8
  Refill reminders: score 1: number analyzed (Participants) | 459
  Refill reminders: score 1 | 27.2
  Refill reminders: score 2: number analyzed (Participants) | 459
  Refill reminders: score 2 | 21.6
  Refill reminders: score 3: number analyzed (Participants) | 459
  Refill reminders: score 3 | 1.1
  Refill reminders: score 4: number analyzed (Participants) | 459
  Refill reminders: score 4 | 50.1
  Newsletters: score 1: number analyzed (Participants) | 460
  Newsletters: score 1 | 15.7
  Newsletters: score 2: number analyzed (Participants) | 460
  Newsletters: score 2 | 19.8
  Newsletters: score 3: number analyzed (Participants) | 460
  Newsletters: score 3 | 1.3
  Newsletters: score 4: number analyzed (Participants) | 460
  Newsletters: score 4 | 63.3
  Reimbursement support: score 1: number analyzed (Participants) | 456
  Reimbursement support: score 1 | 6.8
  Reimbursement support: score 2: number analyzed (Participants) | 456
  Reimbursement support: score 2 | 7.7
  Reimbursement support: score 3: number analyzed (Participants) | 456
  Reimbursement support: score 3 | 1.5
  Reimbursement support: score 4: number analyzed (Participants) | 456
  Reimbursement support: score 4 | 84.0
  Financial assistance: score 1: number analyzed (Participants) | 460
  Financial assistance: score 1 | 4.3
  Financial assistance: score 2: number analyzed (Participants) | 460
  Financial assistance: score 2 | 4.6
  Financial assistance: score 3: number analyzed (Participants) | 460
  Financial assistance: score 3 | 1.3
  Financial assistance: score 4: number analyzed (Participants) | 460
  Financial assistance: score 4 | 89.8
  Other educational materials: score 1: number analyzed (Participants) | 462
  Other educational materials: score 1 | 15.2
  Other educational materials: score 2: number analyzed (Participants) | 462
  Other educational materials: score 2 | 26.4
  Other educational materials: score 3: number analyzed (Participants) | 462
  Other educational materials: score 3 | 0.6
  Other educational materials: score 4: number analyzed (Participants) | 462
  Other educational materials: score 4 | 57.8
  Collection/disposal of sharps container: score 1: number analyzed (Participants) | 456
  Collection/disposal of sharps container: score 1 | 30.0
  Collection/disposal of sharps container: score 2: number analyzed (Participants) | 456
  Collection/disposal of sharps container: score 2 | 23.0
  Collection/disposal of sharps container: score 3: number analyzed (Participants) | 456
  Collection/disposal of sharps container: score 3 | 2.9
  Collection/disposal of sharps container: score 4: number analyzed (Participants) | 456
  Collection/disposal of sharps container: score 4 | 44.1
  Starter pack: score 1: number analyzed (Participants) | 436
  Starter pack: score 1 | 44.5
  Starter pack: score 2: number analyzed (Participants) | 436
  Starter pack: score 2 | 32.6
  Starter pack: score 3: number analyzed (Participants) | 436
  Starter pack: score 3 | 1.4
  Starter pack: score 4: number analyzed (Participants) | 436
  Starter pack: score 4 | 21.6

25. Other Pre Specified Outcome: PSP Satisfaction Questionnaire Responses at Week 24
Description: as for outcome 24
Time Frame: Week 24
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User
Number analyzed (Participants) | 405
percentage of participants
  Relieves my daily burden: score 1: number analyzed (Participants) | 392
  Relieves my daily burden: score 1 | 22.2
  Relieves my daily burden: score 2: number analyzed (Participants) | 392
  Relieves my daily burden: score 2 | 34.9
  Relieves my daily burden: score 3: number analyzed (Participants) | 392
  Relieves my daily burden: score 3 | 15.6
  Relieves my daily burden: score 4: number analyzed (Participants) | 392
  Relieves my daily burden: score 4 | 27.3
  Is always there for me: score 1: number analyzed (Participants) | 391
  Is always there for me: score 1 | 28.9
  Is always there for me: score 2: number analyzed (Participants) | 391
  Is always there for me: score 2 | 38.1
  Is always there for me: score 3: number analyzed (Participants) | 391
  Is always there for me: score 3 | 11.3
  Is always there for me: score 4: number analyzed (Participants) | 391
  Is always there for me: score 4 | 21.7
  Offers real added value service: score 1: number analyzed (Participants) | 387
  Offers real added value service: score 1 | 27.1
  Offers real added value service: score 2: number analyzed (Participants) | 387
  Offers real added value service: score 2 | 39.0
  Offers real added value service: score 3: number analyzed (Participants) | 387
  Offers real added value service: score 3 | 8.5
  Offers real added value service: score 4: number analyzed (Participants) | 387
  Offers real added value service: score 4 | 25.3
  Is exceptional: score 1: number analyzed (Participants) | 389
  Is exceptional: score 1 | 22.9
  Is exceptional: score 2: number analyzed (Participants) | 389
  Is exceptional: score 2 | 43.4
  Is exceptional: score 3: number analyzed (Participants) | 389
  Is exceptional: score 3 | 10.8
  Is exceptional: score 4: number analyzed (Participants) | 389
  Is exceptional: score 4 | 22.9
  PSP in total: score 1: number analyzed (Participants) | 403
  PSP in total: score 1 | 33.5
  PSP in total: score 2: number analyzed (Participants) | 403
  PSP in total: score 2 | 36.7
  PSP in total: score 3: number analyzed (Participants) | 403
  PSP in total: score 3 | 1.5
  PSP in total: score 4: number analyzed (Participants) | 403
  PSP in total: score 4 | 28.3
  Call center/hotline: score 1: number analyzed (Participants) | 400
  Call center/hotline: score 1 | 28.8
  Call center/hotline: score 2: number analyzed (Participants) | 400
  Call center/hotline: score 2 | 27.5
  Call center/hotline: score 3: number analyzed (Participants) | 400
  Call center/hotline: score 3 | 1.8
  Call center/hotline: score 4: number analyzed (Participants) | 400
  Call center/hotline: score 4 | 42.0
  Educational materials about life with RA: score 1 | 31.9
  Educational materials about life with RA: score 2 | 45.7
  Educational materials about life with RA: score 3 | 1.5
  Educational materials about life with RA: score 4 | 21.0
  Educational materials about adalimumab: score 1: number analyzed (Participants) | 399
  Educational materials about adalimumab: score 1 | 34.6
  Educational materials about adalimumab: score 2: number analyzed (Participants) | 399
  Educational materials about adalimumab: score 2 | 42.6
  Educational materials about adalimumab: score 3: number analyzed (Participants) | 399
  Educational materials about adalimumab: score 3 | 0.8
  Educational materials about adalimumab: score 4: number analyzed (Participants) | 399
  Educational materials about adalimumab: score 4 | 22.1
  Injection guide: score 1: number analyzed (Participants) | 403
  Injection guide: score 1 | 44.9
  Injection guide: score 2: number analyzed (Participants) | 403
  Injection guide: score 2 | 39.0
  Injection guide: score 3: number analyzed (Participants) | 403
  Injection guide: score 3 | 0.2
  Injection guide: score 4: number analyzed (Participants) | 403
  Injection guide: score 4 | 15.9
  Nursing services: score 1: number analyzed (Participants) | 400
  Nursing services: score 1 | 27.8
  Nursing services: score 2: number analyzed (Participants) | 400
  Nursing services: score 2 | 16.3
  Nursing services: score 3: number analyzed (Participants) | 400
  Nursing services: score 3 | 1.3
  Nursing services: score 4: number analyzed (Participants) | 400
  Nursing services: score 4 | 54.8
  Email contact: score 1: number analyzed (Participants) | 397
  Email contact: score 1 | 7.6
  Email contact: score 2: number analyzed (Participants) | 397
  Email contact: score 2 | 10.3
  Email contact: score 3: number analyzed (Participants) | 397
  Email contact: score 3 | 1.5
  Email contact: score 4: number analyzed (Participants) | 397
  Email contact: score 4 | 80.6
  Refill reminders: score 1: number analyzed (Participants) | 402
  Refill reminders: score 1 | 26.4
  Refill reminders: score 2: number analyzed (Participants) | 402
  Refill reminders: score 2 | 18.7
  Refill reminders: score 3: number analyzed (Participants) | 402
  Refill reminders: score 3 | 0.2
  Refill reminders: score 4: number analyzed (Participants) | 402
  Refill reminders: score 4 | 54.7
  Newsletters: score 1: number analyzed (Participants) | 396
  Newsletters: score 1 | 11.1
  Newsletters: score 2: number analyzed (Participants) | 396
  Newsletters: score 2 | 22.0
  Newsletters: score 3: number analyzed (Participants) | 396
  Newsletters: score 3 | 2.0
  Newsletters: score 4: number analyzed (Participants) | 396
  Newsletters: score 4 | 64.9
  Reimbursement support: score 1: number analyzed (Participants) | 396
  Reimbursement support: score 1 | 7.1
  Reimbursement support: score 2: number analyzed (Participants) | 396
  Reimbursement support: score 2 | 7.6
  Reimbursement support: score 3: number analyzed (Participants) | 396
  Reimbursement support: score 3 | 0.5
  Reimbursement support: score 4: number analyzed (Participants) | 396
  Reimbursement support: score 4 | 84.8
  Financial assistance: score 1: number analyzed (Participants) | 396
  Financial assistance: score 1 | 4.8
  Financial assistance: score 2: number analyzed (Participants) | 396
  Financial assistance: score 2 | 3.8
  Financial assistance: score 3: number analyzed (Participants) | 396
  Financial assistance: score 3 | 0.8
  Financial assistance: score 4: number analyzed (Participants) | 396
  Financial assistance: score 4 | 90.7
  Other educational materials: score 1: number analyzed (Participants) | 399
  Other educational materials: score 1 | 12.5
  Other educational materials: score 2: number analyzed (Participants) | 399
  Other educational materials: score 2 | 25.8
  Other educational materials: score 3: number analyzed (Participants) | 399
  Other educational materials: score 3 | 0.8
  Other educational materials: score 4: number analyzed (Participants) | 399
  Other educational materials: score 4 | 60.9
  Collection/disposal of sharps container: score 1: number analyzed (Participants) | 398
  Collection/disposal of sharps container: score 1 | 29.1
  Collection/disposal of sharps container: score 2: number analyzed (Participants) | 398
  Collection/disposal of sharps container: score 2 | 22.9
  Collection/disposal of sharps container: score 3: number analyzed (Participants) | 398
  Collection/disposal of sharps container: score 3 | 1.0
  Collection/disposal of sharps container: score 4: number analyzed (Participants) | 398
  Collection/disposal of sharps container: score 4 | 47.0
  Starter pack: score 1: number analyzed (Participants) | 2
  Starter pack: score 1 | 0
  Starter pack: score 2: number analyzed (Participants) | 2
  Starter pack: score 2 | 50.0
  Starter pack: score 3: number analyzed (Participants) | 2
  Starter pack: score 3 | 0
  Starter pack: score 4: number analyzed (Participants) | 2
  Starter pack: score 4 | 50.0

26. Other Pre Specified Outcome: PSP Satisfaction Questionnaire Responses at Week 52
Description: as for outcome 24
Time Frame: Week 52
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User
Number analyzed (Participants) | 346
percentage of participants
  Relieves my daily burden: score 1: number analyzed (Participants) | 336
  Relieves my daily burden: score 1 | 21.7
  Relieves my daily burden: score 2: number analyzed (Participants) | 336
  Relieves my daily burden: score 2 | 32.4
  Relieves my daily burden: score 3: number analyzed (Participants) | 336
  Relieves my daily burden: score 3 | 12.5
  Relieves my daily burden: score 4: number analyzed (Participants) | 336
  Relieves my daily burden: score 4 | 33.3
  Is always there for me: score 1: number analyzed (Participants) | 335
  Is always there for me: score 1 | 28.1
  Is always there for me: score 2: number analyzed (Participants) | 335
  Is always there for me: score 2 | 37.6
  Is always there for me: score 3: number analyzed (Participants) | 335
  Is always there for me: score 3 | 8.4
  Is always there for me: score 4: number analyzed (Participants) | 335
  Is always there for me: score 4 | 26.0
  Offers real added value service: score 1: number analyzed (Participants) | 335
  Offers real added value service: score 1 | 25.4
  Offers real added value service: score 2: number analyzed (Participants) | 335
  Offers real added value service: score 2 | 39.1
  Offers real added value service: score 3: number analyzed (Participants) | 335
  Offers real added value service: score 3 | 9.6
  Offers real added value service: score 4: number analyzed (Participants) | 335
  Offers real added value service: score 4 | 26.0
  Is exceptional: score 1: number analyzed (Participants) | 334
  Is exceptional: score 1 | 21.6
  Is exceptional: score 2: number analyzed (Participants) | 334
  Is exceptional: score 2 | 42.2
  Is exceptional: score 3: number analyzed (Participants) | 334
  Is exceptional: score 3 | 9.6
  Is exceptional: score 4: number analyzed (Participants) | 334
  Is exceptional: score 4 | 26.6
  PSP in total: score 1: number analyzed (Participants) | 339
  PSP in total: score 1 | 33.3
  PSP in total: score 2: number analyzed (Participants) | 339
  PSP in total: score 2 | 36.6
  PSP in total: score 3: number analyzed (Participants) | 339
  PSP in total: score 3 | 1.2
  PSP in total: score 4: number analyzed (Participants) | 339
  PSP in total: score 4 | 28.9
  Call center/hotline: score 1: number analyzed (Participants) | 338
  Call center/hotline: score 1 | 27.2
  Call center/hotline: score 2: number analyzed (Participants) | 338
  Call center/hotline: score 2 | 25.4
  Call center/hotline: score 3: number analyzed (Participants) | 338
  Call center/hotline: score 3 | 1.5
  Call center/hotline: score 4: number analyzed (Participants) | 338
  Call center/hotline: score 4 | 45.9
  Educational materials about life with RA: score 1 | 33.2
  Educational materials about life with RA: score 2 | 41.3
  Educational materials about life with RA: score 3 | 0.9
  Educational materials about life with RA: score 4 | 24.6
  Educational materials about adalimumab: score 1: number analyzed (Participants) | 344
  Educational materials about adalimumab: score 1 | 33.4
  Educational materials about adalimumab: score 2: number analyzed (Participants) | 344
  Educational materials about adalimumab: score 2 | 41.9
  Educational materials about adalimumab: score 3: number analyzed (Participants) | 344
  Educational materials about adalimumab: score 3 | 1.2
  Educational materials about adalimumab: score 4: number analyzed (Participants) | 344
  Educational materials about adalimumab: score 4 | 23.5
  Injection guide: score 1: number analyzed (Participants) | 342
  Injection guide: score 1 | 38.6
  Injection guide: score 2: number analyzed (Participants) | 342
  Injection guide: score 2 | 37.1
  Injection guide: score 3: number analyzed (Participants) | 342
  Injection guide: score 3 | 0.6
  Injection guide: score 4: number analyzed (Participants) | 342
  Injection guide: score 4 | 23.7
  Nursing services: score 1: number analyzed (Participants) | 340
  Nursing services: score 1 | 22.9
  Nursing services: score 2: number analyzed (Participants) | 340
  Nursing services: score 2 | 15.9
  Nursing services: score 3: number analyzed (Participants) | 340
  Nursing services: score 3 | 1.2
  Nursing services: score 4: number analyzed (Participants) | 340
  Nursing services: score 4 | 60.0
  Email contact: score 1: number analyzed (Participants) | 336
  Email contact: score 1 | 5.4
  Email contact: score 2: number analyzed (Participants) | 336
  Email contact: score 2 | 10.1
  Email contact: score 3: number analyzed (Participants) | 336
  Email contact: score 3 | 0.9
  Email contact: score 4: number analyzed (Participants) | 336
  Email contact: score 4 | 83.6
  Refill reminders: score 1: number analyzed (Participants) | 343
  Refill reminders: score 1 | 20.4
  Refill reminders: score 2: number analyzed (Participants) | 343
  Refill reminders: score 2 | 17.5
  Refill reminders: score 3: number analyzed (Participants) | 343
  Refill reminders: score 3 | 1.5
  Refill reminders: score 4: number analyzed (Participants) | 343
  Refill reminders: score 4 | 60.6
  Newsletters: score 1: number analyzed (Participants) | 339
  Newsletters: score 1 | 13.3
  Newsletters: score 2: number analyzed (Participants) | 339
  Newsletters: score 2 | 20.9
  Newsletters: score 3: number analyzed (Participants) | 339
  Newsletters: score 3 | 1.8
  Newsletters: score 4: number analyzed (Participants) | 339
  Newsletters: score 4 | 64.0
  Reimbursement support: score 1: number analyzed (Participants) | 341
  Reimbursement support: score 1 | 6.5
  Reimbursement support: score 2: number analyzed (Participants) | 341
  Reimbursement support: score 2 | 7.3
  Reimbursement support: score 3: number analyzed (Participants) | 341
  Reimbursement support: score 3 | 0.9
  Reimbursement support: score 4: number analyzed (Participants) | 341
  Reimbursement support: score 4 | 85.3
  Financial assistance: score 1: number analyzed (Participants) | 338
  Financial assistance: score 1 | 4.1
  Financial assistance: score 2: number analyzed (Participants) | 338
  Financial assistance: score 2 | 5.0
  Financial assistance: score 3: number analyzed (Participants) | 338
  Financial assistance: score 3 | 1.5
  Financial assistance: score 4: number analyzed (Participants) | 338
  Financial assistance: score 4 | 89.3
  Other educational materials: score 1: number analyzed (Participants) | 337
  Other educational materials: score 1 | 9.5
  Other educational materials: score 2: number analyzed (Participants) | 337
  Other educational materials: score 2 | 26.4
  Other educational materials: score 3: number analyzed (Participants) | 337
  Other educational materials: score 3 | 1.2
  Other educational materials: score 4: number analyzed (Participants) | 337
  Other educational materials: score 4 | 62.9
  Collection/disposal of sharps container: score 1: number analyzed (Participants) | 343
  Collection/disposal of sharps container: score 1 | 28.3
  Collection/disposal of sharps container: score 2: number analyzed (Participants) | 343
  Collection/disposal of sharps container: score 2 | 19.8
  Collection/disposal of sharps container: score 3: number analyzed (Participants) | 343
  Collection/disposal of sharps container: score 3 | 2.0
  Collection/disposal of sharps container: score 4: number analyzed (Participants) | 343
  Collection/disposal of sharps container: score 4 | 49.9

27. Other Pre Specified Outcome: PSP Satisfaction Questionnaire Responses at Week 78
Description: as for outcome 24
Time Frame: Week 78
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Participants With RA Receiving Adalimumab: PSP User
Number analyzed (Participants) | 337
percentage of participants
  Relieves my daily burden: score 1: number analyzed (Participants) | 334
  Relieves my daily burden: score 1 | 22.2
  Relieves my daily burden: score 2: number analyzed (Participants) | 334
  Relieves my daily burden: score 2 | 32.9
  Relieves my daily burden: score 3: number analyzed (Participants) | 334
  Relieves my daily burden: score 3 | 14.1
  Relieves my daily burden: score 4: number analyzed (Participants) | 334
  Relieves my daily burden: score 4 | 30.8
  Is always there for me: score 1: number analyzed (Participants) | 334
  Is always there for me: score 1 | 29.9
  Is always there for me: score 2: number analyzed (Participants) | 334
  Is always there for me: score 2 | 38.3
  Is always there for me: score 3: number analyzed (Participants) | 334
  Is always there for me: score 3 | 7.8
  Is always there for me: score 4: number analyzed (Participants) | 334
  Is always there for me: score 4 | 24.0
  Offers real added value service: score 1: number analyzed (Participants) | 330
  Offers real added value service: score 1 | 25.2
  Offers real added value service: score 2: number analyzed (Participants) | 330
  Offers real added value service: score 2 | 42.1
  Offers real added value service: score 3: number analyzed (Participants) | 330
  Offers real added value service: score 3 | 7.9
  Offers real added value service: score 4: number analyzed (Participants) | 330
  Offers real added value service: score 4 | 24.8
  Is exceptional: score 1: number analyzed (Participants) | 333
  Is exceptional: score 1 | 22.2
  Is exceptional: score 2: number analyzed (Participants) | 333
  Is exceptional: score 2 | 42.0
  Is exceptional: score 3: number analyzed (Participants) | 333
  Is exceptional: score 3 | 9.3
  Is exceptional: score 4: number analyzed (Participants) | 333
  Is exceptional: score 4 | 26.4
  PSP in total: score 1: number analyzed (Participants) | 336
  PSP in total: score 1 | 34.2
  PSP in total: score 2: number analyzed (Participants) | 336
  PSP in total: score 2 | 35.7
  PSP in total: score 3: number analyzed (Participants) | 336
  PSP in total: score 3 | 1.5
  PSP in total: score 4: number analyzed (Participants) | 336
  PSP in total: score 4 | 28.6
  Call center/hotline: score 1: number analyzed (Participants) | 334
  Call center/hotline: score 1 | 27.8
  Call center/hotline: score 2: number analyzed (Participants) | 334
  Call center/hotline: score 2 | 22.2
  Call center/hotline: score 3: number analyzed (Participants) | 334
  Call center/hotline: score 3 | 1.8
  Call center/hotline: score 4: number analyzed (Participants) | 334
  Call center/hotline: score 4 | 48.2
  Educational materials about life with RA: score 1 | 30.3
  Educational materials about life with RA: score 2 | 46.3
  Educational materials about life with RA: score 3 | 1.2
  Educational materials about life with RA: score 4 | 22.3
  Educational materials about adalimumab: score 1: number analyzed (Participants) | 334
  Educational materials about adalimumab: score 1 | 30.5
  Educational materials about adalimumab: score 2: number analyzed (Participants) | 334
  Educational materials about adalimumab: score 2 | 46.1
  Educational materials about adalimumab: score 3: number analyzed (Participants) | 334
  Educational materials about adalimumab: score 3 | 0.9
  Educational materials about adalimumab: score 4: number analyzed (Participants) | 334
  Educational materials about adalimumab: score 4 | 22.5
  Injection guide: score 1: number analyzed (Participants) | 333
  Injection guide: score 1 | 42.0
  Injection guide: score 2: number analyzed (Participants) | 333
  Injection guide: score 2 | 36.6
  Injection guide: score 3: number analyzed (Participants) | 333
  Injection guide: score 3 | 0.6
  Injection guide: score 4: number analyzed (Participants) | 333
  Injection guide: score 4 | 20.7
  Nursing services: score 1: number analyzed (Participants) | 332
  Nursing services: score 1 | 22.6
  Nursing services: score 2: number analyzed (Participants) | 332
  Nursing services: score 2 | 15.7
  Nursing services: score 3: number analyzed (Participants) | 332
  Nursing services: score 3 | 0.6
  Nursing services: score 4: number analyzed (Participants) | 332
  Nursing services: score 4 | 61.1
  Email contact: score 1: number analyzed (Participants) | 326
  Email contact: score 1 | 6.7
  Email contact: score 2: number analyzed (Participants) | 326
  Email contact: score 2 | 9.8
  Email contact: score 3: number analyzed (Participants) | 326
  Email contact: score 3 | 0.6
  Email contact: score 4: number analyzed (Participants) | 326
  Email contact: score 4 | 82.8
  Refill reminders: score 1: number analyzed (Participants) | 326
  Refill reminders: score 1 | 25.5
  Refill reminders: score 2: number analyzed (Participants) | 326
  Refill reminders: score 2 | 16.6
  Refill reminders: score 3: number analyzed (Participants) | 326
  Refill reminders: score 3 | 1.2
  Refill reminders: score 4: number analyzed (Participants) | 326
  Refill reminders: score 4 | 56.7
  Newsletters: score 1: number analyzed (Participants) | 327
  Newsletters: score 1 | 11.6
  Newsletters: score 2: number analyzed (Participants) | 327
  Newsletters: score 2 | 19.6
  Newsletters: score 3: number analyzed (Participants) | 327
  Newsletters: score 3 | 1.8
  Newsletters: score 4: number analyzed (Participants) | 327
  Newsletters: score 4 | 67.0
  Reimbursement support: score 1: number analyzed (Participants) | 326
  Reimbursement support: score 1 | 6.1
  Reimbursement support: score 2: number analyzed (Participants) | 326
  Reimbursement support: score 2 | 7.4
  Reimbursement support: score 3: number analyzed (Participants) | 326
  Reimbursement support: score 3 | 0.9
  Reimbursement support: score 4: number analyzed (Participants) | 326
  Reimbursement support: score 4 | 85.6
  Financial assistance: score 1: number analyzed (Participants) | 324
  Financial assistance: score 1 | 4.0
  Financial assistance: score 2: number analyzed (Participants) | 324
  Financial assistance: score 2 | 5.2
  Financial assistance: score 3: number analyzed (Participants) | 324
  Financial assistance: score 3 | 0.9
  Financial assistance: score 4: number analyzed (Participants) | 324
  Financial assistance: score 4 | 89.8
  Other educational materials: score 1: number analyzed (Participants) | 325
  Other educational materials: score 1 | 12.3
  Other educational materials: score 2: number analyzed (Participants) | 325
  Other educational materials: score 2 | 24.9
  Other educational materials: score 3: number analyzed (Participants) | 325
  Other educational materials: score 3 | 0.6
  Other educational materials: score 4: number analyzed (Participants) | 325
  Other educational materials: score 4 | 62.2
  Collection/disposal of sharps container: score 1: number analyzed (Participants) | 329
  Collection/disposal of sharps container: score 1 | 31.6
  Collection/disposal of sharps container: score 2: number analyzed (Participants) | 329
  Collection/disposal of sharps container: score 2 | 19.8
  Collection/disposal of sharps container: score 3: number analyzed (Participants) | 329
  Collection/disposal of sharps container: score 3 | 2.1
  Collection/disposal of sharps container: score 4: number analyzed (Participants) | 329
  Collection/disposal of sharps container: score 4 | 46.5

ADVERSE EVENTS:
Time Frame: Baseline through Week 78 or early termination
Description: All treatment-emergent serious adverse events (AEs), AEs leading to premature discontinuation from the study, and non-serious AEs of malignancy in patients 30 years of age and younger were collected and are presented. Spontaneously reported non-serious treatment-emergent AEs were also included.
Arm/Group | Participants With RA Receiving Adalimumab
Serious Adverse Events (participants affected / at risk) | 97/1025
Other Adverse Events (participants affected / at risk) | 95/1025
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With RA Receiving Adalimumab (N=1025)
HAEMORRHAGIC DISORDER (Blood and lymphatic system disorders) | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2
ANGINA PECTORIS (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 2
GOITRE (Endocrine disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
DIVERTICULUM (Gastrointestinal disorders) | 1
OESOPHAGEAL HAEMORRHAGE (Gastrointestinal disorders) | 1
PROTEIN-LOSING GASTROENTEROPATHY (Gastrointestinal disorders) | 1
RECTAL PROLAPSE (Gastrointestinal disorders) | 1
DEVICE DAMAGE (General disorders) | 1
MEDICAL DEVICE PAIN (General disorders) | 1
NODULE (General disorders) | 1
PYREXIA (General disorders) | 2
BILE DUCT STONE (Hepatobiliary disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1
APPENDICITIS (Infections and infestations) | 2
ARTHRITIS BACTERIAL (Infections and infestations) | 1
BRONCHIOLITIS (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
CHRONIC TONSILLITIS (Infections and infestations) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1
DIVERTICULITIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
KIDNEY INFECTION (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
MENINGITIS STREPTOCOCCAL (Infections and infestations) | 1
MYCOBACTERIUM MARINUM INFECTION (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 9
SALMONELLOSIS (Infections and infestations) | 1
SALPINGO-OOPHORITIS (Infections and infestations) | 2
SOFT TISSUE INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 2
UROSEPSIS (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 1
WHIPPLE'S DISEASE (Infections and infestations) | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
WOUND (Injury, poisoning and procedural complications) | 1
OBESITY (Metabolism and nutrition disorders) | 2
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 2
MONARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 5
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 8
RHEUMATOID NODULE (Musculoskeletal and connective tissue disorders) | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
DEMYELINATION (Nervous system disorders) | 1
HYPOTONIA (Nervous system disorders) | 1
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 1
SCIATICA (Nervous system disorders) | 1
ANXIETY (Psychiatric disorders) | 1
MAJOR DEPRESSION (Psychiatric disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 1
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
HYPERTENSION (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With RA Receiving Adalimumab (N=1025)
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 2
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1
PALPITATIONS (Cardiac disorders) | 1
TINNITUS (Ear and labyrinth disorders) | 2
VERTIGO (Ear and labyrinth disorders) | 2
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 1
BLEPHARITIS (Eye disorders) | 1
CATARACT (Eye disorders) | 1
KERATITIS (Eye disorders) | 1
VISION BLURRED (Eye disorders) | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 2
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 4
ODYNOPHAGIA (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
ADVERSE DRUG REACTION (General disorders) | 2
ASTHENIA (General disorders) | 5
CHEST PAIN (General disorders) | 1
DEVICE MATERIAL ISSUE (General disorders) | 1
FATIGUE (General disorders) | 3
INFLUENZA LIKE ILLNESS (General disorders) | 1
INJECTION SITE PAIN (General disorders) | 2
INJECTION SITE RASH (General disorders) | 1
INJECTION SITE REACTION (General disorders) | 4
MALAISE (General disorders) | 2
DRUG HYPERSENSITIVITY (Immune system disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 2
ARTHRITIS INFECTIVE (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 2
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
EYE INFECTION (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 2
GENITAL INFECTION FUNGAL (Infections and infestations) | 1
HELICOBACTER INFECTION (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 1
INFECTION SUSCEPTIBILITY INCREASED (Infections and infestations) | 2
INFLUENZA (Infections and infestations) | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
NASOPHARYNGITIS (Infections and infestations) | 1
PERIODONTITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 2
PYELONEPHRITIS (Infections and infestations) | 1
RASH PUSTULAR (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
RHINITIS (Infections and infestations) | 1
TOOTH ABSCESS (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3
URINARY TRACT INFECTION (Infections and infestations) | 5
WOUND INFECTION (Infections and infestations) | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
BLOOD CHOLESTEROL INCREASED (Investigations) | 1
DRUG SPECIFIC ANTIBODY PRESENT (Investigations) | 1
WEIGHT DECREASED (Investigations) | 2
HYPERALBUMINAEMIA (Metabolism and nutrition disorders) | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 2
ACQUIRED CLAW TOE (Musculoskeletal and connective tissue disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1
MUSCLE FATIGUE (Musculoskeletal and connective tissue disorders) | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 4
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1
BENIGN NEOPLASM OF PROSTATE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
DIZZINESS (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 7
MIGRAINE (Nervous system disorders) | 1
PINEAL GLAND CYST (Nervous system disorders) | 1
SCIATICA (Nervous system disorders) | 1
SENSORY LOSS (Nervous system disorders) | 1
ANXIETY (Psychiatric disorders) | 2
DEPRESSION (Psychiatric disorders) | 2
INSOMNIA (Psychiatric disorders) | 1
IRRITABILITY (Psychiatric disorders) | 1
LOSS OF LIBIDO (Psychiatric disorders) | 1
SLEEP DISORDER (Psychiatric disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 2
DERMATITIS PSORIASIFORM (Skin and subcutaneous tissue disorders) | 3
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 3
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 8
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1
ROSACEA (Skin and subcutaneous tissue disorders) | 1
SKIN REACTION (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 2
FLUSHING (Vascular disorders) | 1
HAEMORRHAGE (Vascular disorders) | 1
HOT FLUSH (Vascular disorders) | 1
HYPERTENSION (Vascular disorders) | 4
PHLEBITIS (Vascular disorders) | 1
VASCULITIS (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.